CLINICAL TRIAL: NCT06669949
Title: Natural History and Phenotypic Spectrum of Sphingosine Phosphate Lyase Insufficiency Syndrome (SPLIS)
Brief Title: Natural History of Sphingosine Phosphate Lyase Insufficiency Syndrome (SPLIS)
Acronym: SPLIS-HIS
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-37968; R01HD113778 (NIH)
Record Dates: First submitted 2024-10-26; First posted 2024-11-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Sphingosine Phosphate Lyase Insufficiency Syndrome (SPLIS)
Keywords: sphingosine phosphate lyase; SGPL1; sphingolipidosis; steroid-resistant nephrotic syndrome; neurological defect; sphingolipid; nephrotic syndrome; primary adrenal insufficiency; primary immunodeficiency; Charcot-Marie-Tooth Disease; hypothyroidism; ichthyosis; sphingosine phosphate lyase insufficiency syndrome; RENI syndrome; NPHS14
MeSH Terms: conditions — Sphingolipidoses; Nephrotic Syndrome; Addison Disease; Primary Immunodeficiency Diseases; Charcot-Marie-Tooth Disease; Hypothyroidism; Ichthyosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood will be collected for plasma and peripheral blood mononuclear cells. Urine and stool samples will be collected. Leftover material not used in clinical testing will be retained for future research use. Leftover skin biopsy material or fibroblasts derived from skin biopsies obtained as part of medical care may be used to create a cell line that will be analyzed and stored in a specimen bank at University of California San Francisco.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with sphingosine phosphate lyase insufficiency syndrome: Individuals diagnosed with sphingosine phosphate lyase insufficiency syndrome based on genetic testing that confirms bi-allelic pathogenic variants in the SGPL1 gene
  Interventions: Other: no intervention
- Parents of individuals with sphingosine phosphate lyase insufficiency syndrome: Parents of individuals diagnosed with sphingosine phosphate lyase insufficiency syndrome based on genetic testing that confirms bi-allelic pathogenic variants in the SGPL1 gene
  Interventions: Other: no intervention
- age and gender-matched controls: The investigators will attempt to collect biological specimens from individuals closely matched to SPLIS patient cohort by age and gender. This group may include siblings, cousins, and unrelated healthy children and adults.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No interventions are involved in this observational study.

SUMMARY:
This is a prospective longitudinal natural history study with a retrospective cross-sectional arm aimed at determining the natural history of sphingosine phosphate lyase insufficiency syndrome (SPLIS), a recently recognized inborn error of metabolism. The central hypothesis is that age of onset, other disease features, and disease biomarkers will be predictive of quality of life (QOL) and survival in SPLIS patients.

DETAILED DESCRIPTION:
The main purpose of the study is to characterize the natural history of sphingosine phosphate lyase insufficiency syndrome (SPLIS) including the full spectrum of presentations (clinical, biochemical, radiological and pathological) and their change (progression or improvement) over time by collecting and analyzing data from prospective assessments on patients with SPLIS over a three-year time period and retrospective chart review of treatment history. By necessity, the investigators will also endeavor to explore the range of medical treatments and interventions currently being used in the care of SPLIS patients and their impact on the natural history of SPLIS. A retrospective arm will collect data on patients who are deceased and/or who are willing to share medical data but unwilling to participate in the prospective arm of the study.

The secondary objective of the study is to establish a set of biomarkers including plasma sphingosine-1-phosphate (S1P) and absolute lymphocyte count (ALC) that may aid in:

* Characterizing distinct phenotypic subgroups of SPLIS patients within the larger SPLIS population
* Predicting the change (progression or improvement) in symptoms of SPLIS patients over time

The exploratory objectives of the study are to explore the potential of plasma sphingolipids other than S1P, urinary sphingolipids including S1P, and immunological markers including cytokines and T cell subsets to serve as disease biomarkers. A SPLIS multi-domain responder index (MDRI) will be developed. Induced pluripotent stem cells derived from peripheral blood mononuclear cells and/or skin fibroblasts will be generated as a research tool.

ELIGIBILITY:
All identified patients with SPLIS diagnosed by genetic criteria are eligible for enrollment in this study, regardless of baseline demographic, biochemical or metabolic features and regardless of interventions such as vitamin B6 supplementation, dialysis or kidney transplantation at time of enrollment. This study may include siblings of index SPLIS cases if the sibling has been genetically confirmed to have SPLIS, regardless of whether they have active disease at the time of enrollment. Data from deceased SPLIS patients will also be collected.

Inclusion Criteria:

Potential subjects fulfilling the following criteria will be eligible to participate in this study:

1. Living or deceased patients diagnosed with SPLIS based on

   1. harbor biallelic pathogenic variant (PV) or likely PV (LPV) in the SGPL1 gene, regardless of phenotype OR
   2. harbor nucleotide changes in both SGPL1 alleles, regardless of variant classification, if they also have one of the following: b1) exhibit at least 1 phenotypic feature of SPLIS (nephrosis, endocrine defect, ichthyosis, neuropathy, male gonadal dysgenesis, lymphopenia) b2) have evidence from biochemical or molecular data (such as enzyme expression or activity in skin fibroblasts) that indicate a possible loss of function in the S1P lyase (SPL) protein b3) are a sibling of a subject with nucleotide changes in both alleles of SGPL1 and at least 1 phenotypic feature of SPLIS
2. Informed consent and (if appropriate) assent for living subjects. For deceased subjects, the Principal Investigator (PI) will be responsible for ensuring that all requirements have been met in regard to the relevant local laws and regulations. Parents of participating SPLIS patients may be included as controls.

Exclusion Criteria:

Subjects with SPLIS (or their parents) who are currently using or have a history of using an investigational agent in the last 30 days with the exception of off-label use of medications will be excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SPLIS is a genetic disorder caused by recessive mutations in SGPL1. The study population includes individuals with confirmed bi-allelic mutations in SGPL1, regardless of age, gender, disease manifestations, or treatments received. Some patients with SPLIS will have kidney failure, adrenal insufficiency and/or neurological problems. Parents, family members and unrelated healthy individuals enrolled during routine health appointments, elective surgical procedures and other medical interactions will be included as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 years
  The primary outcome of this study is survival (age at death).
Height | 3 years
  Standing height, sitting height and knee height in centimeters will be performed by stadiometer over time.
Weight | 3 years
  Weight in kilograms will be measured by weight scale over time.
Head circumference | 3 years
  Head circumference in centimeters will be measured by insertion tape over time.
Triceps skin fold measurement | 3 years
  Skin fold in centimeters by skinfold calipers will be measured at the mid-triceps region over time.
Subscapular skin fold measurement | 3 years
  Skin fold in centimeters by skinfold calipers will be measured at the subscapular region over time.
Upper arm muscle circumference | 3 years
  Upper arm muscle circumference in centimeters will be measured using a tape measure over time.
Sitting height | 3 years
  Sitting height in centimeters will be measured using a stadiometer over time.
Knee height | 3 years
  Knee height in centimeters will be measured using a knee height caliper over time.
Tibial length | 3 years
  Tibial length in centimeters will be measured using a tape measure over time.
Nutritional intake assessment | 3 years
  A questionnaire assessing 24-hour recall of nutritional intake will be performed using using a 3-day food log. The information will be assessed using the online Automated Self-Administered 24-Hour Dietary Recall (ASA24) tool. The nutritional intake assessment will additionally include information on emesis and stool consistently using the Bristol Stool Chart.
Retinal condition | 3 years
  Retinal condition will be assessed using a non-dilated eye exam.
Skin condition | 3 years
  Appearance of acanthoses, ichthyosis, skin barrier function will be performed by a Tewameter instrument over time.
Charcot Marie Tooth Neuropathy Score (CMTNS) | 3 years
  Charcot Marie Tooth neuropathy scores are made up of nine assessments, including three symptoms, four signs, and two neurophysiology items tested by nerve conduction study. Each assessment is scored on a scale of 0-4, with higher scores indicating greater impairment.
Abdominal ultrasound | At baseline
  An abdominal ultrasound will be performed to evaluate kidney and adrenal gland structure.
Audiology testing | 3 years
  Hearing will be tested over time using standard audiology testing methods.
Cognitive function | 3 years
  Cognitive function will be tested using the Vineland Adaptive Behavior Scales developmental test. The Vineland scales consist of questions about communication, daily living, socialization, and motor skills, and questions are targeted to age and developmental stage, rated on a scale of 0 (not able to perform behavior) to 2 (completely able to perform behavior). Cognitive testing will additionally include the Leiter-3.0, a nonverbal intelligence test designed to assess the cognitive abilities of individuals, primarily those who may have language or communication barriers. The exact interpretation of these scores is typically done by a trained psychologist or clinician, who will consider the test results in context with other information to provide a comprehensive assessment.
Tanner stage | 3 years
  Sexual maturity will be determined by Tanner stage during physical exam. As Tanner stages move 1 through 5 to characterize the development of secondary sexual characteristics for males and females.
Proteinuria | 3 years
  Proteinuria will be measured as urine albumin/creatinine ratio (ACR) determined with a 24 hour urine collection.
Serum creatinine | 3 years
  Serum creatinine will be measured in mg/dL and used to determine estimated glomerular filtration rate (eGFR) in units of (mL/min/1.73m2) over time.
Thyroid function | 3 years
  Free thyroxine (T4) and thyroid stimulating hormone by blood sample will be measured over time.
Cortisol | 3 years
  Morning cortisol level in micrograms/deciliter by blood sample will be measured over time.
Adrenocorticotropin hormone (ACTH) | 3 years
  ACTH in picograms per milliliter will be measured by blood sample over time.
Renin | 3 years
  Blood renin measured in nanograms/milliliter/hour will be measured over time.
Testosterone | 3 years
  Testosterone will be measured in nanograms/deciliter by blood sample over time.
Estradiol | 3 years
  Estradiol will be measured in picograms per milliliter by blood sample over time.
Anti-mullerian hormone (AMH) | 3 years
  Anti-mullerian hormone will be measured in nanograms/milliliter by blood sample over time.
Inhibin B | 3 years
  Inhibin B will be measured in picograms per milliliter by blood sample over time.
Follicle stimulating hormone (FSH) | 3 years
  Follicle stimulating hormone will be measured in milli international units per milliliter (mIU/ml) by blood sample over time.
Luteinizing hormone (LH) | 3 years
  Luteinizing hormone will be measured in international units per liter (IU/L) by blood sample over time.
Insulin-like growth factor 1 (IGF-1) | 3 years
  IGF-1 will be measured in nanograms/mL by blood over time.
Blood glucose | 3 years
  Blood glucose will be measured in milligrams per deciliter by blood sample over time.
Serum sodium | 3 years
  Serum sodium will be measured in milliequivalents per liter by blood sample over time.
Serum potassium | 3 years
  Serum potassium will be measured in milliequivalents per liter by blood sample over time.
Serum chloride | 3 years
  Serum chloride will be measured in milliequivalents per liter by blood sample over time.
Serum carbon dioxide (CO2) | 3 years
  Serum CO2 will be measured in milliequivalents per liter by blood sample over time.
Complete blood count | 3 years
  A complete automated blood count will be performed by blood sample over time.
Serum immunoglobulins | 3 years
  Serum immunoglobulins (IgG, IgA, IgM) will be measured by blood sample over time.
Antibodies to vaccine | At baseline
  Antibodies to childhood vaccinations by blood sample will be measured.
Blood urea nitrogen (BUN) | 3 years
  BUN will be measured in mg/dL by blood sample over time.
Patient journey questionnaire | At baseline
  A patient journey questionnaire capturing timing of disease feature onset and progression will be completed by the patient/family.
Pediatric Quality of Life (PedsQL) Questionnaires | At baseline
  PedsQL is a validated and standardized questionnaire capturing information on pediatric quality of life. The study will use 4 modules to capture various patients: End Stage Renal Disease Module, Family Impact Module, Generic Core Scales, and the Infant Scales. A higher score indicates a higher quality of life.
Cholesterol panel | 3 years
  A cholesterol profile including high, low, and very low density lipoprotein (HDL, LDL, VLDL) and total cholesterol by blood sample will be measured.
Pre- and Post-Kidney Transplant Questionnaire | 3 years
  A questionnaire capturing pre- and post-kidney transplant clinical information will be completed by the patient's physician (if applicable).
Echocardiography | 3 years
  A standard cardiac ultrasound will be performed by a pediatric cardiologist to track SPLIS-related cardiovascular changes or abnormalities including left and chamber sizes and masses, Doppler measurements, and aortic diameter.
Edema-Related Quality of Life | 3 years
  As SPLIS patients often experience edema as a result of kidney failure, PREPARE-NS is a questionnaire that will be used to gage how kidney failure symptoms like edema alter a patient's quality of living.
Patient-Reported Outcomes Measurement Information System (PROMIS) | 3 years
  PROMIS assesses quality of life in several domains including physical functioning, mental health, social functioning, pain, sleep, fatigue, cognitive functioning, emotional distress, and ability to participate in social roles and activities. A higher score indicates a high quality of life.
Cystatin C | 3 years
  Cystatin C will be measured in milligrams per liter (mg/L) or micrograms per milliliter (µg/mL) using a blood sample to assess kidney function.
Urine specific gravity | 3 years
  Urine specific gravity will be measured using a urine sample, a unitless measure comparing the ratio of the density of urine to water, providing information about the kidney's ability to concentrate or dilute urine.
Skin Barrier Function uingTewameter, Sebumeter, and Corneometer | 3 years
  Skin barrier function will be measured using a device called a Multi-Probe Adapter-5 (MPA5) manufactured by Courage + Khazaka, which uses a tewameter probe (measuring transepidermal water loss), a sebumeter (measuring skin sebum), and a corneometer (measuring skin hydration).

SECONDARY OUTCOMES:
Blood sphingolipid levels | 3 years
  Blood levels of sphingosine-1-phosphate, dihydrosphingosine-1-phosphate, sphingosine, dihydrosphingosine and ceramides will be measured by blood sample using tandem mass spectrometry over time and reported in micromolarity units.
Urine sphingolipid levels | 3 years
  Urine levels of sphingosine-1-phosphate, dihydrosphingosine-1-phosphate, sphingosine, dihydrosphingosine and ceramides will be measured in a 24 hour urine collection using tandem mass spectrometry over time and reported in micromolarity units.
Sphingolipid levels from skin biopsy | 1-6 weeks
  Skin fibroblast sphingolipid levels will be collected using skin biopsy, and compared by liquid chromatography/mass spectrometry in medium containing various therapeutic agents. This test will be performed to characterize the response to interventions in fibroblasts.
Sphingosine phosphate lyase (SPL) enzyme activity from skin biopsy | 1-6 weeks
  Skin fibroblast SPL activity levels will be measured by skin biopsy using liquid chromatography/mass spectrometry in response to interventions in fibroblasts.

OTHER OUTCOMES:
Lymphocyte subsets | 3 years
  CD3, CD4, CD8, CD20, CD56/16 positive cells and recent thymic emigrants representing lymphocyte subsets in the peripheral blood will be measured over time by blood sample and reported as absolute numbers of cells/mm^3.
Multi-Domain Responder Index | 3 years
  Patients will be asked to review their symptoms every 6 months, while their parents (when applicable) will be asked to review their own, and recall their family history of relevant symptoms. The multidomain responder index is a scoring system that tailors a score to the patient's worst symptoms, which will be created as a result of symptom tracking. Scoring arbitrarily starts at 0 on the first measurement and may stay at 0 on subsequent exams (no change over time), increase to +1 (improvement over time), or decrease to -1 (worsening over time). This will be tested for ability to measure overall patient status over time.
Pyridoxal 5'-phosphate (PLP) | 3 years
  PLP, the active form of vitamin B6, will be measured by blood sample over time if patients are planning to or have initiated cofactor supplementation with pyridoxine.
Occult blood presence by stool sample | 3 years
  Occult blood will be tested by stool sample only if gastrointestinal symptoms are present. This test is done through a chemical detection of heme.
Stool fat by stool sample | 3 years
  Stool fat will be tested by stool sample only if gastrointestinal symptoms are present.
Stool reducing substances by stool sample | 3 years
  Stool reducing substances will be tested by stool sample only if gastrointestinal symptoms are present using qualitative chromaticity - the process of identifying the hue or color of stool (brown, green, yellow, black, or red) to detect an underlying gut health abnormality. Brown is normal, while a change to any other color suggests a deviation from normal.
Calprotectin by stool sample | 3 years
  Calprotectin will be tested by stool sample only if gastrointestinal symptoms are present, using quantitative chemiluminescent immunoassay - a technique that replies on the use of light to detect the concentration of calprotectin in stool. Moderate (50-120 ug/g) to high (>120 ug/g) levels of calprotectin indicate moderate to high levels of gut inflammation.
Gut microbiome by stool sample | 3 years
  Gut microbiome analysis will be performed using DNA extraction and 16s gene sequencing from a stool sample over time to assess the microorganism composition of the intestines, affecting gut health.
Skin fibroblasts for neural reprogramming | At baseline
  Skin fibroblasts will be obtained through a skin biopsy and subsequently reprogrammed to differentiate into neurons. This process will be used for basic science research.
Skin fibroblasts for induced pluripotent stem cells (iPSCs) | At baseline
  Skin fibroblasts or peripheral blood mononuclear cells will be obtained through a skin biopsy and subsequently reprogrammed to become iPSCs. This process will be used for basic science research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Julie D Saba, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller N, Midgley J, Khalid E, Lesmana H, Mathew G, Mincham C, Teig N, Khan Z, Khosla I, Mehr S, Guran T, Buder K, Xu H, Alhasan K, Buyukyilmaz G, Weaver N, Saba JD. Factors influencing survival in sphingosine phosphate lyase insufficiency syndrome: a retrospective cross-sectional natural history study of 76 patients. Orphanet J Rare Dis. 2024 Sep 27;19(1):355. doi: 10.1186/s13023-024-03311-w. PMID 39334450
- [Background] Lovric S, Goncalves S, Gee HY, Oskouian B, Srinivas H, Choi WI, Shril S, Ashraf S, Tan W, Rao J, Airik M, Schapiro D, Braun DA, Sadowski CE, Widmeier E, Jobst-Schwan T, Schmidt JM, Girik V, Capitani G, Suh JH, Lachaussee N, Arrondel C, Patat J, Gribouval O, Furlano M, Boyer O, Schmitt A, Vuiblet V, Hashmi S, Wilcken R, Bernier FP, Innes AM, Parboosingh JS, Lamont RE, Midgley JP, Wright N, Majewski J, Zenker M, Schaefer F, Kuss N, Greil J, Giese T, Schwarz K, Catheline V, Schanze D, Franke I, Sznajer Y, Truant AS, Adams B, Desir J, Biemann R, Pei Y, Ars E, Lloberas N, Madrid A, Dharnidharka VR, Connolly AM, Willing MC, Cooper MA, Lifton RP, Simons M, Riezman H, Antignac C, Saba JD, Hildebrandt F. Mutations in sphingosine-1-phosphate lyase cause nephrosis with ichthyosis and adrenal insufficiency. J Clin Invest. 2017 Mar 1;127(3):912-928. doi: 10.1172/JCI89626. Epub 2017 Feb 6. PMID 28165339
- [Background] Prasad R, Hadjidemetriou I, Maharaj A, Meimaridou E, Buonocore F, Saleem M, Hurcombe J, Bierzynska A, Barbagelata E, Bergada I, Cassinelli H, Das U, Krone R, Hacihamdioglu B, Sari E, Yesilkaya E, Storr HL, Clemente M, Fernandez-Cancio M, Camats N, Ram N, Achermann JC, Van Veldhoven PP, Guasti L, Braslavsky D, Guran T, Metherell LA. Sphingosine-1-phosphate lyase mutations cause primary adrenal insufficiency and steroid-resistant nephrotic syndrome. J Clin Invest. 2017 Mar 1;127(3):942-953. doi: 10.1172/JCI90171. Epub 2017 Feb 6. PMID 28165343
- [Background] Weaver KN, Sullivan B, Hildebrandt F, Strober J, Cooper M, Prasad R, Saba J. Sphingosine Phosphate Lyase Insufficiency Syndrome. 2020 Oct 15. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK562988/ PMID 33074640
- [Background] Zhao P, Liu ID, Hodgin JB, Benke PI, Selva J, Torta F, Wenk MR, Endrizzi JA, West O, Ou W, Tang E, Goh DL, Tay SK, Yap HK, Loh A, Weaver N, Sullivan B, Larson A, Cooper MA, Alhasan K, Alangari AA, Salim S, Gumus E, Chen K, Zenker M, Hildebrandt F, Saba JD. Responsiveness of sphingosine phosphate lyase insufficiency syndrome to vitamin B6 cofactor supplementation. J Inherit Metab Dis. 2020 Sep;43(5):1131-1142. doi: 10.1002/jimd.12238. Epub 2020 May 4. PMID 32233035
- [Background] Martin KW, Weaver N, Alhasan K, Gumus E, Sullivan BR, Zenker M, Hildebrandt F, Saba JD. MRI Spectrum of Brain Involvement in Sphingosine-1-Phosphate Lyase Insufficiency Syndrome. AJNR Am J Neuroradiol. 2020 Oct;41(10):1943-1948. doi: 10.3174/ajnr.A6746. Epub 2020 Aug 27. PMID 32855188
- [Background] Zhao P, Tassew GB, Lee JY, Oskouian B, Munoz DP, Hodgin JB, Watson GL, Tang F, Wang JY, Luo J, Yang Y, King S, Krauss RM, Keller N, Saba JD. Efficacy of AAV9-mediated SGPL1 gene transfer in a mouse model of S1P lyase insufficiency syndrome. JCI Insight. 2021 Apr 22;6(8):e145936. doi: 10.1172/jci.insight.145936. PMID 33755599